CLINICAL TRIAL: NCT01456260
Title: A Phase 3, Multicenter, Single-blind, AG-1749-controlled, Parallel-group, Long-term Extension Study to Evaluate the Safety and Efficacy of TAK-438 (10 mg or 20 mg, Orally, Once Daily) for the Prevention of Recurrent Gastric or Duodenal Ulcers During Long-term Therapy of Non-steroidal Anti-inflammatory Drug (NSAID)
Brief Title: Long-term Extension Study of TAK-438 for the Prevention of Recurrent Gastric or Duodenal Ulcers During Therapy of Non-steroidal Anti-inflammatory Drug (NSAID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TAK-438/OCT-301; U1111-1123-8762 (Registry Identifier: WHO); JapicCTI-111611 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-16; First posted 2011-10-20 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Gastric Ulcers; Duodenal Ulcers
Keywords: Drug Therapy
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-438 10 mg QD (Experimental)
  Interventions: Drug: TAK-438; Drug: Placebo
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438; Drug: Placebo
- Lansoprazole 15 mg QD (Active Comparator)
  Interventions: Drug: Lansoprazole; Drug: Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 10 mg tablets, orally, once daily for 28-80 weeks.
  Arms: TAK-438 10 mg QD
Drug: Placebo — Lansoprazole placebo matching capsules, orally, once daily for 28-80 weeks.
  Arms: TAK-438 10 mg QD
Drug: TAK-438 — TAK-438 20 mg tablets, orally, once daily for 28-80 weeks.
  Arms: TAK-438 20 mg QD
Drug: Placebo — Lansoprazole placebo-matching capsules, orally, once daily for 28-80 weeks.
  Arms: TAK-438 20 mg QD
Drug: Lansoprazole — Lansoprazole 15 mg capsules, orally, once daily for 28-80 weeks.
  Other Names: AG-1749
  Arms: Lansoprazole 15 mg QD
Drug: Placebo — TAK-438 placebo-matching tablets, orally, once daily for 28-80 weeks.
  Arms: Lansoprazole 15 mg QD

SUMMARY:
The purpose of this study is to evaluate the safety of TAK-438, once daily (QD), during long-term concomitant non-steroidal anti-inflammatory drug (NSAID) therapy in patients with a history of gastric or duodenal ulcer who require long-term therapy of NSAID.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who require continuous NSAID therapy during the treatment period with the study drug
2. Participants who have completed the preceding study
3. Outpatient (including inpatient for examinations)

Exclusion Criteria:

1. Participants deemed to be ineligible to participate in the study by the principal investigator or investigator due to the occurrence of adverse events in the preceding study
2. Participants who are scheduled to change the type and dosage regimen of NSAID
3. Participants with ulcers or bleeding in stomach or duodenum, endoscopically confirmed during the preceding study
4. Participants with small intestine bleeding, large intestine bleeding, or gastrointestinal bleeding of unknown etiology
5. Participants who have a history of surgery which affects gastric acid secretion (e.g., resection of upper gastrointestinal tract, vagotomy) or who are scheduled to undergo such surgery
6. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders
7. Participants with a previous or current history of aspirin-induced asthma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2011-09; Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 80 weeks.
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through the last visit of study.

SECONDARY OUTCOMES:
Change from baseline in Laboratory values | Up to 80 weeks.
Change from baseline in Electrocardiograms | Up to 80 weeks.
Change from baseline in Vital signs | Up to 80 weeks.
Change from baseline in Serum gastrin | Up to 80 weeks.
Change from baseline in Pepsinogen I and II | Up to 80 weeks.
Recurrence rate of gastric or duodenal ulcer | Up to 80 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (97):
- Japan (97):
  - Kasugai-shi, Aichi-ken
  - Nagoya, Aichi-ken
  - Seto-shi, Aichi-ken
  - Akita, Akita
  - Funabashi-shi, Chiba
  - Ichihara-shi, Chiba
  - Nagareyama-shi, Chiba
  - Matsuyama, Ehime
  - Niihama-shi, Ehime
  - Saijo-shi, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Itoshima-shi, Fukuoka
  - Kitakyusyu-shi, Fukuoka
  - Munakata-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Tagawa-shi, Fukuoka
  - Yukuhashi-shi, Fukuoka
  - Fukushima, Fukushima
  - Koriyama-shi, Fukushima
  - Mebashi-shi, Gunma
  - Takasaki-shi, Gunma
  - Fukuyama-shi, Hiroshima
  - Hatsukaichi-shi, Hiroshima
  - Higashihirosima-shi, Hiroshima
  - Asahikawa-shi, Hokkaido
  - Hakodate-shi, Hokkaido
  - Obihiro-shi, Hokkaido
  - Sapporo, Hokkaido
  - Sunagawa-shi, Hokkaido
  - Tomakomai-shi, Hokkaido
  - Akashi-shi, Hyōgo
  - Himeji-shi, Hyōgo
  - Itami-shi, Hyōgo
  - Kako-gun, Hyōgo
  - Kato-shi, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya-shi, Hyōgo
  - Higashiibaragi-gun, Ibaragi
  - Koga-shi, Ibaragi
  - Mito, Ibaragi
  - Hakusan-shi, Ishikawa-ken
  - Komatsu-shi, Ishikawa-ken
  - Takamatsu, Kagawa-ken
  - Kamakura-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Uji-shi, Kyoto
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Matsumoto-shi, Nagano
  - Nagano, Nagano
  - Nagasaki, Nagasaki
  - Ikoma-shi, Nara
  - Nara, Nara
  - Nigata-shi, Niigata
  - Beppu-shi, Oita Prefecture
  - Ōita, Oita Prefecture
  - Yuhu-shi, Oita Prefecture
  - Kurashiki-shi, Okayama-ken
  - Higashiosaka-shi, Osaka
  - Moriguchi-shi, Osaka
  - Osaka, Osaka
  - Osakasayama-shi, Osaka
  - Tondabayashi-shi, Osaka
  - Ogi-shi, Saga-ken
  - Ageo-shi, Saitama
  - Hiki-gun, Saitama
  - Kasukabe-shi, Saitama
  - Kumagaya-shi, Saitama
  - Saitama-shi, Saitama
  - Sayama-shi, Saitama
  - Toda-shi, Saitama
  - Tokorozawa-shi, Saitama
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Naruto-shi, Tokushima
  - Adachi-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Hachiouji-shi, Tokyo
  - Koto-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashimurayama-shi, Tokyo
  - Nakano-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Sumida-ku, Tokyo
  - Yonago-shi, Tottori
  - Tonami-shi, Toyama
  - Toyama, Toyama
  - Shimonoseki-shi, Yamaguchi
  - Ube-shi, Yamaguchi

REFERENCES:
- [Derived] Mizokami Y, Oda K, Funao N, Nishimura A, Soen S, Kawai T, Ashida K, Sugano K. Vonoprazan prevents ulcer recurrence during long-term NSAID therapy: randomised, lansoprazole-controlled non-inferiority and single-blind extension study. Gut. 2018 Jun;67(6):1042-1051. doi: 10.1136/gutjnl-2017-314010. Epub 2017 Oct 7. PMID 28988197